CLINICAL TRIAL: NCT07114809
Title: Impact of Anodal tDCS and Virtual Reality on Cognitive Dysfunction in Patients With Multiple Sclerosis: a Protocol of a Double Blind, Randomized, Prospective, Controlled Study.
Brief Title: Impact of Anodal tDCS and Virtual Reality on Cognitive Dysfunction in Patients With Multiple Sclerosis
Acronym: tDCScog
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Policlinico San Martino (Other)
Collaborators: Italian Multiple Sclerosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/R-Multi/034
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Impairment; Multiple Sclerosis
Keywords: Cognitive impairment; Multiple Sclerosis; Exergaiming; Virtual Reality; tDCS
MeSH Terms: conditions — Cognitive Dysfunction; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: double blind, randomized, controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (EG) performing Anodal-tDCS (A-tDCS) and VR (Experimental): EG subjects will undergo a rehabilitative treatment with exergame and concurrent A-tDCS over the left dorsolateral prefrontal cortex.
  Interventions: Device: Experimental group (EG) performing Anodal-tDCS (A-tDCS) and VR
- Control group (CG) performing sham-tDCS (S-tCDS) and VR (Sham Comparator): CG subjects will undergo a rehabilitative treatment with exergame and concurrent S-tDCS over the left dorsolateral prefrontal cortex.
  Interventions: Device: Sham Comparator: Control group (CG) performing sham-tDCS (S-tCDS) and VR

INTERVENTIONS:
Device: Experimental group (EG) performing Anodal-tDCS (A-tDCS) and VR — Patients in the EG group will undergo a simultaneous A-tDCS over the left DLFPC. The tDCS will be delivered by a battery-driven, constant current simulator, two holding bags of plant cellulose (7x5 cm) and two electrodes of conductive silicone. The active (anodal) electrode will be placed by means of a cap on the scalp overlying the left DLPFC (46 Brodmann Area). The reference electrode will be located over the right shoulder. The choice of the left DLPFC as the site of stimulation relies upon the evidence that this region has a critical role in the "top-down" control of the task-relevant stimuli processing (Miller 2001).The DLPFC contributes to increase cognitive control through its connections with the anterior cingulate cortex and has been shown to enhance working memory and executive function. During the cognitive training (on-line procedure), A-tDCS (current of 1,5 mA) will be delivered for 20 minutes, while maintaining the current density (0.06 mA/cm2) below the safety limits.
  Arms: Experimental group (EG) performing Anodal-tDCS (A-tDCS) and VR
Device: Sham Comparator: Control group (CG) performing sham-tDCS (S-tCDS) and VR — CG will receive a S-tDCS over the DLPFC. In the S-tDCS session, the current will be turned off 30 sec after the beginning of the stimulation and turned on for the last 30 sec. By doing this, the patient feels an itching sensation below the electrodes at the beginning and at the end of stimulation, making this condition indistinguishable from the real A-tDCS stimulation. Doing this, all the subjects will be blinded on the type of stimulation. As well as in the EG, CG performs cognitive training including motor and cognitive exergames that incorporate enjoyment, technology, and health care.
  Arms: Control group (CG) performing sham-tDCS (S-tCDS) and VR

SUMMARY:
Cognitive impairment (CI) affects a large amount of patients with Multiple Sclerosis (PwMS) even in the early stages of the disease, increasing the perception of fatigue and compromising the quality of life. Different restorative interventions have been tried in order to alleviate CI, but with limited efficacy .

Transcranial direct current stimulation (tDCS), represents a very promising alternative, or add-on, to the traditional rehabilitative approaches in MS. Notably, other novel technologies, such as Virtual Reality (VR) and Exergame, are emerging as a reinforcing tool to the rehabilitative treatment of PwMS. tDCS and VR can be combined in protocols aimed at achieving a better therapeutic benefit across different neurological diseases (Cassani 2020). The aim of our project is to explore the potential benefits of the simultaneous application of AtDCS and VR in the rehabilitation of cognitive impairment of PwMS. The VR approach will be implemented with a non-immersive VR system (exergames). As a secondary outcome, we wish to verify whether our protocol may extend its benefits over 6 months. Eighty PwMs with CI will be consecutively enrolled. Their cognitive status will be assessed by a neuropsychological battery: the Brief International Cognitive Assessment for MS and the Paced Auditory Serial Addition Test. To be considered cognitively impaired one has to abnormally score on at least two tests. Forty patients will be randomized to the experimental group (EG) or to the control group (CG). All the patients will undergo rehabilitative treatment with exergame (10 sessions for two consecutive weeks, 5 days per week). The EG patients will undergo a concurrent A-tDCS over the left dorsolateral prefrontal cortex, while the CG will receive a sham stimulation (S-tDCS). The patients will be evaluated at baseline, at the end of the treatment, one month and six months later. The statistical analyses will be done using repeated-measures ANOVA. Expected results: we hypothesize that the cognitive performances of both EG and CG groups will show an improvement in the cognitive performances. We will expect, however, a significative difference between the two groups, with patients in the EG group demonstrating better results than the CG group. Finally, we hypothesize the beneficial effects in EG patients will last at least one month after the end of the experiment.

DETAILED DESCRIPTION:
To achieve our aims, we planned a double-blind, randomized, prospective, controlled study. To this purpose, we will recruit 80 MS subjects affected by cognitive impairment (CI). Patients will be selected from outpatients attending the Department of Neurology of ASL3 Genoa and the Neurorehabilitation unit of IRCCS Ospedale Policlinico San Martino, Genoa. The participants will be randomly assigned to two groups, 40 in the experimental group (EG), 40 in the control group (CG), matched for demographic data (gender, age), EDSS and disease duration. All subjects will undergo a cognitive training by means of the exergames system (10 sessions, one hour per session, 5 days per week, for two consecutive weeks). Patients in the EG group will undergo a simultaneous A-tDCS over the left DLFPC, while CG will receive a S-tDCS over the same area. The tDCS will be delivered by a battery-driven, constant current simulator with a LCD touch screen (HDC progr), a portable stimulator (HDC stim), two holding bags of plant cellulose (7x5 cm) and two electrodes of conductive silicone. The active (anodal) electrode will be placed by means of a cap on the scalp overlying the left DLPFC (46 Brodmann Area). The reference electrode will be located over the right shoulder. The choice of the left DLPFC as the site of stimulation relies upon the evidence that this region has a critical role in the "top-down" control of the task-relevant stimuli processing .

In addition, in tasks where a cognitive conflict arises, the DLPFC contributes to increased cognitive control through its connections with the anterior cingulate cortex . Finally A-tDCS of the DLPFC has been shown to enhance working memory and executive function in healthy subjects as well as in PwMS . An electroconductive gel will be applied under the electrodes in order to reduce contact impedance. Impedance will be constantly kept below 5 kOhm. Only the tDCS investigators will be aware of the type of stimulation, while the patients and the neuropsychological assessors will be blind as to the nature of the project. During the exergames training (on-line procedure), A-tDCS (current of 1,5 mA) will be delivered for 20 minutes, while maintaining the current density (0.06 mA/ cm2) below the safety limits . In the StDCS session (20 minutes) the current will be turned off 30 sec after the beginning of the stimulation and turned on for the last 30 sec. By doing this, the patient feels an itching sensation below the electrodes at the beginning and at the end of stimulation, making this condition indistinguishable from the real (anodic) stimulation. Doing this, all the subjects will be blinded on the type of stimulation (anodal or sham). All the patients will participate to the cognitive training by means of exergames, which includes motor and cognitive tasks that incorporate enjoyment, technology, and health care.

ELIGIBILITY:
Inclusion Criteria:

1. MS diagnosis according to McDonald's criteria (McDonald 2017);
2. age between 18 and 60 (to avoid participants with possible CI due to aging); 3) disability score ≤7.5 at the Expanded Disability Status Scale (EDSS, Kurtzke 1983).

Exclusion Criteria:

1. subjects affected by major psychiatric disorders
2. epilepsy
3. previous brain surgery
4. MS relapse requiring steroid therapy in the previous two months
5. bilateral visual acuity < 6/10

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Revised Brief Visuo-Spatial Memory test (BVMT-R) | The patients will be evaluated at baseline, up to two weeks, one month and six months later
  Part of the BICAMS test. minimum score 0 (poor performance) maximum score 12 (normal performance)
Symbol digit modalities test (SDMT) | The patients will be evaluated at baseline, up to two weeks, one month and six months later.
  Part of the BICAMS test. minimum score 0 (poor performance), maximum score 120 (normal performance)
California Verbal Learning test II edition (CVLT-II) | The patients will be evaluated at baseline, up to two weeks, one month and six months later
  Part of the BICAMS test. Minimum score 0 (poor performance), maximum score 80 (normal performance)
Paced Auditory Serial Addition Task 3" and 2" intervals (PASAT) | The patients will be evaluated at baseline, up to two weeks, one month and six months later
  A neuropsychological test widely utilized for the cognitive assessment in PwMS. Minimum score 0 (poor performance) maximum score 60 (normal performance)

SECONDARY OUTCOMES:
Multiple Sclerosis Quality of life (MSQoL) | The patients will be evaluated at baseline, up to two weeks, one month and six months later
  Self-reported measures of quality of life in people with Multiple Sclerosis. Minimum score 0 (poor performance), Maximum score 100 (normal performance)
Beck depression inventory scale (BDI) | The patients will be evaluated at baseline, up to two weeks, one month and six months later
  Self-reported measures of mood (depression). Minimum score 0 (poor performance), maximum score 63 (normal performance)
Fatigue Severity Scale (FSS) | The patients will be evaluated at baseline, up to two weeks, one month and six months later
  Self-reported measures of fatigue in people with Multiple Sclerosis. Minimum score 9, maximum score 63. (Mean score ≥ 4: indicative of clinically significant fatigue. Mean score < 4: fatigue not considered clinically significant.)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mori, MD, PhD, Principal Investigator — Ospedale Policlinico San Martino IRCCS
Locations (3):
- Italy (3):
  - Azienda Sanitaria Genovese, Genova, Italy
  - Ospedale Policlinico San Martino - IRCCS, Genova, Italy
  - Italian multiple sclerosis foundation, Genova, Italy

IPD SHARING:
Plan to Share IPD: No
At this time, individual participant data (IPD) will not be shared due to concerns regarding patient confidentiality and the challenges of fully anonymizing sensitive clinical and neuropsychological data. In addition, data sharing is not currently covered by participant informed consent and would require additional ethical and regulatory approvals to ensure compliance with privacy laws and institutional policies.

REFERENCES:
- [Background] Laver KE, George S, Thomas S, Deutsch JE, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2015 Feb 12;2015(2):CD008349. doi: 10.1002/14651858.CD008349.pub3. PMID 25927099
- [Background] Cassani R, Novak GS, Falk TH, Oliveira AA. Virtual reality and non-invasive brain stimulation for rehabilitation applications: a systematic review. J Neuroeng Rehabil. 2020 Oct 31;17(1):147. doi: 10.1186/s12984-020-00780-5. PMID 33129331
- [Background] Solari A, Filippini G, Mendozzi L, Ghezzi A, Cifani S, Barbieri E, Baldini S, Salmaggi A, Mantia LL, Farinotti M, Caputo D, Mosconi P. Validation of Italian multiple sclerosis quality of life 54 questionnaire. J Neurol Neurosurg Psychiatry. 1999 Aug;67(2):158-62. doi: 10.1136/jnnp.67.2.158. PMID 10406981
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Charvet L, Shaw M, Dobbs B, Frontario A, Sherman K, Bikson M, Datta A, Krupp L, Zeinapour E, Kasschau M. Remotely Supervised Transcranial Direct Current Stimulation Increases the Benefit of At-Home Cognitive Training in Multiple Sclerosis. Neuromodulation. 2018 Jun;21(4):383-389. doi: 10.1111/ner.12583. Epub 2017 Feb 22. PMID 28225155
- [Background] Mattioli F, Bellomi F, Stampatori C, Capra R, Miniussi C. Neuroenhancement through cognitive training and anodal tDCS in multiple sclerosis. Mult Scler. 2016 Feb;22(2):222-30. doi: 10.1177/1352458515587597. Epub 2015 May 26. PMID 26014600
- [Background] Filippi M, Riccitelli G, Mattioli F, Capra R, Stampatori C, Pagani E, Valsasina P, Copetti M, Falini A, Comi G, Rocca MA. Multiple sclerosis: effects of cognitive rehabilitation on structural and functional MR imaging measures--an explorative study. Radiology. 2012 Mar;262(3):932-40. doi: 10.1148/radiol.11111299. PMID 22357892
- [Background] Mainero C, Caramia F, Pozzilli C, Pisani A, Pestalozza I, Borriello G, Bozzao L, Pantano P. fMRI evidence of brain reorganization during attention and memory tasks in multiple sclerosis. Neuroimage. 2004 Mar;21(3):858-67. doi: 10.1016/j.neuroimage.2003.10.004. PMID 15006652
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Hiew S, Nguemeni C, Zeller D. Efficacy of transcranial direct current stimulation in people with multiple sclerosis: a review. Eur J Neurol. 2022 Feb;29(2):648-664. doi: 10.1111/ene.15163. Epub 2021 Nov 19. PMID 34725881
- [Background] Grigorescu C, Chalah MA, Lefaucheur JP, Kumpfel T, Padberg F, Ayache SS, Palm U. Effects of Transcranial Direct Current Stimulation on Information Processing Speed, Working Memory, Attention, and Social Cognition in Multiple Sclerosis. Front Neurol. 2020 Oct 15;11:545377. doi: 10.3389/fneur.2020.545377. eCollection 2020. PMID 33178103
- [Background] Nascimento AS, Fagundes CV, Mendes FADS, Leal JC. Effectiveness of Virtual Reality Rehabilitation in Persons with Multiple Sclerosis: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Mult Scler Relat Disord. 2021 Sep;54:103128. doi: 10.1016/j.msard.2021.103128. Epub 2021 Jul 9. PMID 34280679
- [Background] Seeley WW, Menon V, Schatzberg AF, Keller J, Glover GH, Kenna H, Reiss AL, Greicius MD. Dissociable intrinsic connectivity networks for salience processing and executive control. J Neurosci. 2007 Feb 28;27(9):2349-56. doi: 10.1523/JNEUROSCI.5587-06.2007. PMID 17329432
- [Background] McNicholas N, O'Connell K, Yap SM, Killeen RP, Hutchinson M, McGuigan C. Cognitive dysfunction in early multiple sclerosis: a review. QJM. 2018 Jun 1;111(6):359-364. doi: 10.1093/qjmed/hcx070. PMID 28371862
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] De Giglio L, De Luca F, Prosperini L, Borriello G, Bianchi V, Pantano P, Pozzilli C. A low-cost cognitive rehabilitation with a commercial video game improves sustained attention and executive functions in multiple sclerosis: a pilot study. Neurorehabil Neural Repair. 2015 Jun;29(5):453-61. doi: 10.1177/1545968314554623. Epub 2014 Nov 14. PMID 25398725
- [Background] Dardiotis E, Nousia A, Siokas V, Tsouris Z, Andravizou A, Mentis AA, Florou D, Messinis L, Nasios G. Efficacy of computer-based cognitive training in neuropsychological performance of patients with multiple sclerosis: A systematic review and meta-analysis. Mult Scler Relat Disord. 2018 Feb;20:58-66. doi: 10.1016/j.msard.2017.12.017. Epub 2017 Dec 24. PMID 29306740
- [Background] Manuli A, Maggio MG, Tripoli D, Gulli M, Cannavo A, La Rosa G, Sciarrone F, Avena G, Calabro RS. Patients' perspective and usability of innovation technology in a new rehabilitation pathway: An exploratory study in patients with multiple sclerosis. Mult Scler Relat Disord. 2020 Sep;44:102312. doi: 10.1016/j.msard.2020.102312. Epub 2020 Jun 18. PMID 32585618
- [Background] Lang N, Siebner HR, Ward NS, Lee L, Nitsche MA, Paulus W, Rothwell JC, Lemon RN, Frackowiak RS. How does transcranial DC stimulation of the primary motor cortex alter regional neuronal activity in the human brain? Eur J Neurosci. 2005 Jul;22(2):495-504. doi: 10.1111/j.1460-9568.2005.04233.x. PMID 16045502
- [Background] Taylor MJ, Griffin M. The use of gaming technology for rehabilitation in people with multiple sclerosis. Mult Scler. 2015 Apr;21(4):355-71. doi: 10.1177/1352458514563593. Epub 2014 Dec 22. PMID 25533296
- [Derived] Vestito L, Schenone C, Casazza F, Modenesi R, Iandolino A, Matichecchia MG, Saez LM, Botto M, Ponzano M, Gazzola P, Grange E, Brichetto G, Bandini F, Trompetto C, Mori L. Impact of anodal tDCS and virtual reality on cognitive dysfunction in patients with Multiple Sclerosis: Protocol of a double blind, randomized, prospective, controlled study. PLoS One. 2025 Dec 4;20(12):e0337405. doi: 10.1371/journal.pone.0337405. eCollection 2025. PMID 41343474